CLINICAL TRIAL: NCT05811572
Title: Investigation of Pelvic Floor Muscle Strength in Women With Low Back Pain
Brief Title: Investigation of Pelvic Floor Muscle Strength in Low Back Pain
Status: Completed | Type: Observational
Sponsor: Gulhan Yilmaz Gokmen (Other)
Responsible Party: Sponsor-Investigator, Gulhan Yilmaz Gokmen, Assistant Professor, Bandırma Onyedi Eylül University
Organization: Bandırma Onyedi Eylül University (Other)
Other Study IDs: 00-2020-0018
Record Dates: First submitted 2023-03-31; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-03

CONDITIONS: Low Back Pain, Mechanical; Pelvic Floor Muscle Weakness; Non-specific Low Back Pain; Disability Physical; Pain
Keywords: Non-specific low back pain; perinometer; Pelvic Floor Muscle; Disability; Pain
MeSH Terms: conditions — Low Back Pain; Pain | interventions — Visual Analog Scale

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With Non-Specific Low Back Pain: pelvic floor muscles measurement with perinometer
  Interventions: Device: measurement of pelvic floor muscle with perinometer
- Without Low Back Pain: pelvic floor muscles measurement with perinometer
  Interventions: Device: measurement of pelvic floor muscle with perinometer

INTERVENTIONS:
Device: measurement of pelvic floor muscle with perinometer — Questions the person's perceptions about low back pain and related disability VAS questions the person's perceptions about low back pain severity
  Other Names: Roland morris disability questionnaire; Visual Analog Scale (VAS)

SUMMARY:
To evaluate the effect of pelvic floor muscle strength on women with non-specific low back pain

ELIGIBILITY:
Inclusion Criteria:

* being a woman
* 18-50 years old
* BMI≤30

For The NSLBP Group:

* diagnosed with non-specific low back pain by a specialist physician,
* have low back pain for at least 3 months,
* have no pain radiating to the leg,
* have low back pain 3 or higher on the visual analog scale (VAS, 0-10 scale)

Exclusion Criteria:

* have a somatic or psychiatric disorder,
* have signs and symptoms associated with other conditions such as nerve root compression (at least 2 of these symptoms: weakness, reflex changes or loss of sensation associated with the same spinal nerve),
* have had previous spinal surgery or are scheduled for surgery,
* Pregnant
* have neurological and pelvic inflammatory diseases

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: Women with and without non-specific low back pain
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
pelvic floor muscle strength | 1 day
  It was done with a manual perinometer. A manometer measuring between 0 and 25 mbar was used. The manometer is connected to the vaginal probe by a plastic, hollow, 75 cm long tube. The diameter of the vaginal probe is 3.5 cm and the length is 15 cm. The vaginal probe is inserted intravaginally to a depth of 5-10 cm. With the person in the supine position, with the knees flexed at 45 degrees, the measurement is made with a perineometer 3 times. For each measurement, the vaginal probe is removed and reinserted intravaginally. Each measurement starts when the indicator part on the manometer is 0 mbar and the patient is asked to tighten the pelvic floor muscles maximally. The average of the three measurements gives the mean pelvic floor muscle strength value.

SECONDARY OUTCOMES:
Roland morris disability questionnaire | 1 day
  First published in 1983 and reviewed in 2000, the Roland-Morris Disability Questionnaire(RMDQ) is designed to assess self-rated physical disability caused by low back pain.There are different questionnaires available, which differ from each other in the number of statements: 24-, 18- and 11-item questionnaires. The score ranges from 0 (no disability) to 24 (max. disability) depending on the questionnaire used.
Visual analog scale | 1 day
  On a 10-centimeter ruler drawn from zero to ten, the individual is asked to mark the most severe pain they have experienced in the last 24 hours. Values of 1-2-3 describe mild pain, values of 4-5-6 describe moderate pain, and 7-8-9-10 describe severe pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Bandırma Onyedi Eylül University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Balıkesir, Turkey (Türkiye)